CLINICAL TRIAL: NCT01123811
Title: An Open-label, Non-randomized Phase II Trial of Cetuximab in Combination With Irinotecan and 5-FU/FA for Patients With Metastatic Gastric Cancer
Brief Title: Efficacy of Cetuximab in Combination With Irinotecan and 5- FU/FA in Treatment of Metastatic Gastric Cancer
Acronym: GC-CIF-2005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: AIO-Studien-gGmbH (Other)
Responsible Party: M Moehler, Johannes Gutenberg University Mainz
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-CIF-2005
Record Dates: First submitted 2010-05-07; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2006-03

CONDITIONS: Adenocarcinoma of Stomach or Esophagogastric Junction
Keywords: adenocarcinoma; gastric cancer; esophagogastric junction cancer
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab IF (Experimental): Treatment with combination of Cetuximab and Irinotecan 5-FU
  Interventions: Drug: Cetuximab IF

INTERVENTIONS:
Drug: Cetuximab IF — Cetuximab loading dose 400 mg/m² weekly dose 250 mg/m² Irinotecan 80 mg/m2 i.v. over 2 hours day 1, 8, 15, 22, 29, 36 Folinic acid 200 mg/m2 over 24 hours day 1, 8, 15, 22, 29, 36 FA will be given as sodium folinate 5-FU 1500 mg/m2 continuous infusion over 24 hours day 1, 8, 15, 22, 29, 36
  Other Names: na-folinat oncofolic

SUMMARY:
Based on the current promising results with irinotecan and cetuximab in patients with recurrent metastatic colorectal cancer, and the excellent results of Irinotecan and 5-FU in gastric cancer , the present clinical study to evaluate the overall response rate, the time to progression and the overall survival of the combined treatment of cetuximab and irinotecan and 5-FU in patients with esophagogastric cancer is urgently needed.

DETAILED DESCRIPTION:
Cetuximab will be analysed with biological markers

ELIGIBILITY:
Inclusion Criteria:

Signed and dated informed consent before the start of specific protocol procedures;

* Histologically proven gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction or Barrett carcinoma (adenocarcinoma of lower oesophagus);
* Measurable metastatic disease according to the RECIST criteria. If locally recurrent disease, it must be associated with at least one measurable lymph node (> 20 mm by CT scan or > 10 mm with spiral CT);
* Age: 18-75 years;
* ECOG Performance Status 0-2
* Life expectancy > 12 weeks;
* Adequate hematological, hepatic and renal functions: ANC

  ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L; hemoglobin ≥ 10g/dl; creatinine ≤ 2 x UNL; total bilirubin ≤ 3 x UNL, ASAT (SGOT) and ALAT (SGPT) ≤ 3 × UNL; in case of liver metastases: total bilirubin ≤ 5 x UNL, ASAT (SGOT) and ALAT (SGPT) ≤ 5 × UNL;
* At least 4 weeks from surgery;
* Recovery from side effects of any prior therapy;
* Able to comply with scheduled assessments and with management of toxicity.
* If of childbearing potential, willingness to use effective contraceptive method for the study duration and 2 months post-dosing.

Exclusion Criteria:

* Other tumor type than adenocarcinoma (e.g., leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix which has been effectively treated. Patients curatively treated and disease free for at least 5 years will be discussed with the sponsor before inclusion;

  * Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol;
  * Any prior palliative chemotherapy, adjuvant (and/or neoadjuvant) chemotherapy or radiotherapy ;
  * Concurrent treatment with any other anti-cancer therapy;
  * Patients with known brain or leptomeningeal metastasis;
  * Hypercalcemia not controlled by bisphosphonates;
  * Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (> hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis;
  * Other serious illness or medical conditions:
* Unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry; congestive heart failure NYHA grade 3 and 4;
* Current history of chronic diarrhea;
* History of significant neurologic or psychiatric disorders including dementia or seizures;
* Active uncontrolled infection;
* Active disseminated intravascular coagulation;
* Other serious underlying medical conditions which could impair the ability of the patient to participate in the study;

  * Known deficit in DPD
  * Contraindications to the use of atropine;
  * Concomitant or within a 4-week period administration of any other experimental drug under investigation;
  * Pregnant or lactating women;
  * Previous exposure to monoclonal antibodies, signal transduction inhibitors or EGFR pathway targeting therapy;
  * Known allergic/hypersensitivity reaction to any of the components of the treatment;
  * Known drug abuse/alcohol abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
objective response rate | 1 month

SECONDARY OUTCOMES:
Progression-free survival | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: M Moehler, Md Ph D, Principal Investigator — Johannes Gutenberg Univetsity
Locations (10):
- Germany (10):
  - Städtische Kliniken Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Klinikum Ludwigsburg, Medizinische Klinik I, Ludwigsburg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Abt. Innere Medizin I, Ulm, Baden-Wurttemberg
  - Klinikum rechts der Isar der technischen Universität München, III. Medizinische Klinik: Hämatologie / Onkologie, München, Bavaria
  - Medizinische Hochschule Hannover, Abteilung Gastroenterologie, Hepatologie und Endokrinologie, Hanover, Lower Saxony
  - Universitätsklinkum Essen, Innere Klinik und Poliklinik - Tumorforschung, Essen, North Rhine-Westphalia
  - Kliniken Essen-Mitte / Evang. Huyssens-Stiftung, Klinik für Innere Medizin I und Internistische Onkologie / Hämatologie, Essen, North Rhine-Westphalia
  - Prosper-Hospital Recklinghausen, Medizinische Klinik I, Recklinghausen, North Rhine-Westphalia
  - Klinikum der Johannes Gutenberg-Universität, I. Medizinische Klinik u. Poliklinik, Mainz, Rhineland-Palatinate
  - Charité - Campus Benjamin Franklin, Medizinische Klinik I, Berlin, State of Berlin